CLINICAL TRIAL: NCT07005700
Title: Development of Rapid Diagnostics for Genetic Disorders in Neonates Using a Novel Targeted Genomic DNA Sequencing Analysis Panel.
Brief Title: Rapid Diagnostics for Genetic Disorders in Neonates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: MedySapiens (Unknown)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director, Neonatal Research Institute, Sharp Mary Birch Hospital for Women and Newborns, Sharp HealthCare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MedySeq
Record Dates: First submitted 2025-04-09; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Acid Base Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Consented, Enrolled (Experimental): All participants who meet inclusion and exclusion criteria and whose parent has provided written informed consent.
  Interventions: Diagnostic Test: Targeted genomic sequencing

INTERVENTIONS:
Diagnostic Test: Targeted genomic sequencing — Single 0.5 mL venous or capillary blood sample.

SUMMARY:
The goal of this study is to test a prototype genomic blood analysis for identifying rare diseases in infants hospitalized in the neonatal intensive care unit (NICU).

The main question it aims to answer is: Does the prototype accurately identify genetic variation(s) associated with an infant's health condition?

Researchers will compare the prototype's gene identification to traditional genome sequencing methods of gene identification.

Participants will be asked to provide a very small (one-tenth of a teaspoon) sample of blood, one-time.

ELIGIBILITY:
Inclusion Criteria: neonates of any gestational age.

* Abnormality in routine neonatal screening test.
* Unexplained neonatal hypotonia or neonate-onset seizures.
* Unexplained and abnormal biochemical laboratory findings.
* Skeletal dysplasia or joint problems.

Exclusion Criteria:

* Parental refusal of consent to participate.
* Provider refusal.
* Any condition that, in the opinion of the investigator, would interfere with interpretation of study results.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Identification of genes associated with congenital diseases | birth through hospital discharge or up to 1 month of age
  A finding that a participant has one of the genes among the 254 included in the targeted gene panel being used. These genes are associated with metabolic, lysosomal storage, immunodeficiency, hemoglobinopathy, and channelopathy diseases, sensorineural hearing loss, and other conditions typically exposed through newborn screening.

CONTACTS AND LOCATIONS:
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim MJ, Kim SY, Lee JS, Kang S, Park LJ, Choi W, Jung JY, Kim T, Park SS, Ko JM, Seong MW, Chae JH. Rapid Targeted Sequencing Using Dried Blood Spot Samples for Patients With Suspected Actionable Genetic Diseases. Ann Lab Med. 2023 May 1;43(3):280-289. doi: 10.3343/alm.2023.43.3.280. Epub 2022 Dec 22. PMID 36544340
- See also: Gene sequencing panel and bioinformatics software being used in the study. — https://medysapiens.com/en/solutions/medycvi